CLINICAL TRIAL: NCT06798545
Title: First-in-human Integrated Endoscopic Ultrasound (EUS) Navigation System Clinical Study
Acronym: EZ-EUS1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IHU Strasbourg (Other)
Collaborators: IRCAD (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 23-002
Record Dates: First submitted 2025-01-21; First posted 2025-01-29 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Diseases
Keywords: endoscopic ultrasound; EUS; navigation; pancreatic disease; training; education; learning curve
MeSH Terms: conditions — Pancreatic Diseases | interventions — Endosonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EUS with EZ-EUS navigation system (Experimental): EUS with the experimental navigation system
  Interventions: Device: endoscopic ultrasound with navigation system
- Standard EUS (No Intervention): EUS in standard condition

INTERVENTIONS:
Device: endoscopic ultrasound with navigation system — Use of the EZ-EUS navigation system during the procedure
  Arms: EUS with EZ-EUS navigation system

SUMMARY:
The complexity of the medical expertise required for endoscopic manipulation and image interpretation complicates the implementation of echo-endoscopy (or EUS for "Endoscopic Ultrasound").

The "EZ-EUS" system is designed to help the operator understand the orientation and the position of the probe tip in the patient. This system offers navigation similar to that of the Global Positioning System (GPS), but for EUS procedures. To achieve this, it uses a 3D model based on scanner imaging data recorded before the procedure.

In this study, the intended purpose of the "EZ-EUS" system is to help echo-endoscopy operators to easily identify and assess the pancreatic gland, and to facilitate the detection of any lesions.

The hypothesis is that, thanks to this tool, procedure times will be shortened, and the pancreas and its lesions will be fully imaged to facilitate their localization and characterization.

DETAILED DESCRIPTION:
Since its inception in the 1980s, the field of endoscopic ultrasound (EUS) has experienced significant expansion and evolution and is now a pivotal component of pancreatobiliary assessment. Proficiency in EUS necessitates a synthesis of cognitive and technical competencies encompassing endoscopic manipulation, image interpretation, and an extensive comprehension of intraabdominal anatomical structures. Acquisition of these competencies is a progressive and highly operator-dependent process, and thereby necessitates an extended learning curve for practitioners.

The American Society for Gastrointestinal Endoscopy (ASGE) has recommended the performance of a minimum of 190 supervised EUS for practicing autonomous EUS. However, the compliance of these parameters does not guarantee competence achievement, and there is a wide variability between endoscopists leading to disparities in the techniques' quality and irregular outcomes.

The "EZ-EUS" system is designed to help the operator understand the orientation and the position of the probe tip in the patient. This system offers navigation similar to that of the Global Positioning System (GPS), but for EUS procedures. To achieve this, it uses a 3D model based on scanner imaging data recorded before the procedure.

In this study, the intended purpose of the "EZ-EUS" system is to assist echo-endoscopy operators in accurately locating the pancreatic gland, conducting a comprehensive evaluation of the region of interest, and facilitating the detection and identification of lesions within it. We hypothesize that this tool will streamline procedure times and enable comprehensive imaging of the pancreas and its lesions, thereby reducing the need for expert guidance for trainees and shortening the EUS learning curve. This study is exploratory, prospective, monocentric and will compare two randomized groups (with and without the EZ-EUS navigation system).

ELIGIBILITY:
Inclusion Criteria:

* Man or woman over the age of 18 years old.
* Patient having a EUS procedure for pancreas study planned within the frame of his or her clinical care.
* Patient whom pre-operative imaging indicates one lesion, a suspicion of lesion, chronic pancreatitis or fatty pancreas.
* Patient with a good definition on the CT scan done within the year to the EUS.
* Patient able to receive and understand information related to the study and give his or her written consent.
* Patient affiliated to the French social security system.

Exclusion Criteria:

* Patient with altered anatomy of the upper digestive tract due to previous surgery.
* Patient with known abnormal anatomy of the upper digestive tract.
* Patient wearing a pacemaker.
* Patients with comorbidities that may increase the risk of perforation.
* Patient presenting, according to the investigator's judgment, a disease which may prevent participation in the procedures provided for by the study.
* Patient with an ASA >3. Patient with ASA=3 must be validated by the Principal
* Investigator (PI).
* Patient unable to tolerate general anesthesia.
* Patient with a body mass index (BMI) < 18,5 and > 40.
* Patient with weight variations >10% between the date on which the CT scan was performed and the date of the procedure.
* Pregnant or lactating patient.
* Patient in exclusion period (determined by a previous or a current study).
* Patient under guardianship or trusteeship.
* Patient under the protection of justice of deprives of liberty.
* Patient in situation of emergency

Perprocedure exclusion criteria

• Patient in need of the balloon during the navigation will be excluded of the study (Experimental group)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the EUS navigation system's procedure duration compared to standard procedure times | 1 day
  Comparison of the examination period duration between the two groups (experimental vs control)

SECONDARY OUTCOMES:
Assessment of the EUS navigation system for patient safety | 1 month
  Rate of adverse events, adverse device effects and complications
Assessment of the system's ease-of-use and technological maturity | 1 day
  Qualitative assessment of the system's ease-of-use and technological maturity using questionnaires. Appropriate statistical test will be used to compare each procedure. Results will be presented numerically and graphically.
Assessment of the EUS navigation system for reliability | 1 day
  Rate of device deficiencies during the procedure
Evaluation of the time required to perform individual step duration | 1 day
  Comparison of the duration of each individual step
Recording of procedure data for offline systeme performance assessment | 1 day
  Collection and prospective review of EUS data, including video and electromagnetic coordinates provided by the sensor
Assessment of the registration method | 1 day
  Quantitative (numerical) assessment of registration accuracy using Target Registration Error (TRE), defined as the distance between the predicted 3D location of an anatomical landmark by the navigation system and its true 3D location

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo SOSA-VALENCIA, MD, Principal Investigator — IHU Strasbourg, HUS
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No